CLINICAL TRIAL: NCT06845293
Title: AO CSH Mainstream Study on Cervical Spine Degeneration
Acronym: CASDEM
Status: Not yet recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASDEM
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cervical Spine Degenerative Disease
Keywords: Cervical Spine Degenerative Disease; prospective multicenter patient cohort; anterior fusion; posterior fusion; Clinical Study Hub

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Adult patients with cervical degenerative diseases undergoing primary anterior and/or posterior cervical fusion will be prospectively enrolled from participating sites.

Patients will be treated and followed up at the participating sites per local standard of care. Several variables related to the patient characteristics and fusion details will be collected. The mainstream study will not collect follow-up (FU) data.

The duration of this patient cohort is currently planned as open ended.

DETAILED DESCRIPTION:
Degeneration of the cervical spine is common and encompasses a wide range of pathologies including spondylosis, central canal and neuroforaminal stenosis, facet arthropathy, and ligamentous hypertrophy. Prevalence of MRI cervical degenerative increases with age. Degenerative changes of cervical intervertebral disc from C2 to C7, including loss of signal intensity, posterior and anterior disc protrusion, narrowing of the disc space, and foraminal stenosis, in 497 asymptomatic subjects using MRI; rates of degenerative changes were 17% in males and 12% in females in their 20s and 86% and 89% in males and females in their 60s, respectively. Ten years later, 223 of the 497 subjects were assessed again (FU rate: 44.9%), and the authors reported an overall rate of degenerative changes of 81%, and 34% of subjects developed clinical symptoms. In a 20-year FU of 193 of the 497 subjects (FU rate: 38.8%), the authors found that degenerative changes have progressed in 95% of the subjects, and gross structural failures like anterior compression of the dura/spinal cord and posterior disc protrusion started in half of the subjects in their 30s, gradually worsened with age, and were detected in > 80% of subjects ≥ 40 years of age.

Degeneration of the cervical spine develops over the time due to structural load, repetitive microtrauma, and age-related changes to the spinal axis. The process typically starts with the intervertebral disc physiology resulting in a loss of the supportive nature of the discs and osteophyte formation, which give rise to spinal canal stenosis and chronic compression of the spinal cord. The structural changes may also lead to hypermobility or spondylolisthesis, which, if unstable, will cause dynamic injuries and repetitive microtrauma to the neural elements. C5-C6 is the most affected level owing to its high mobility and increased weight load.

Patients with cervical degeneration may present with a spectrum of symptoms ranging from generalized neck pain, mechanical or axial neck pain, to debilitating neurologic symptoms such as radiculopathy and myelopathy. Degenerative cervical myelopathy is most worrisome presentation and is the most common nontraumatic spinal cord injury with a wide range of symptoms such as hand numbness and paresthesia, gait impairment, motor weakness of the upper and lower extremities, and bladder and bowel dysfunction. Annual incidence of cervical radiculopathy and myelopathy has been estimated as approximately 83 cases per 100,000 persons and 4 per 100,000 persons.

State of the art of the research field Various treatment algorithms have been proposed to manage cervical degeneration Nonsurgical care including analgesics, chronic pain management physical therapy, supervised exercise and manual therapy, acupuncture, and epidural glucocorticoid injections can provide sufficient relief of chronic neck pain and/or radiculopathy. Surgical treatments are indicated especially in the cases of progressive or significant neurologic symptoms and myelopathy. In the past decades, there is an increase of surgical treatments for cervical degenerative radiculopathy or myelopathy as a result of increased availability of MRI diagnostics, an ageing population, advances in surgical techniques, and easier access to specialist healthcare services.

Surgical approaches for treating cervical degenerative radiculopathy or myelopathy include anterior, posterior, and anteroposterior techniques. The goals of the surgery are to adequately decompress the nerve root or spinal cord and stabilize the spinal column while restoring or maintaining relatively normal spinal alignment. ACDF is a recognized and effective surgical treatment for cervical degenerative disease. In a randomized controlled trial of patients with single-level cervical radiculopathy, ACDF plus physiotherapy showed significant improvement in neck disability, demonstrated by a mean reduction of Neck Disability Index score of 21% (95% confidence interval [CI]: 14 - 28%) after 5 to 8 years, compared with 11% (95% CI: 4 - 18%) in the physiotherapy alone group (p = 0.03). Research is ongoing to identify factors predictive of a good or bad outcome of ACDF and techniques to improve the surgical outcomes.

Patient factors influencing surgical outcomes include bone mineral density, diabetes, smoking, body mass index, vitamin D, and steroid use . Techniques to improve surgical outcomes include alternative to autogenous bone grafts , cage materials/size/height/location (such as polyetheretherketone [PEEK], titanium [Ti], Ti/PEEK combined cages, carbon fiber-reinforced polymers, polymethyl methacrylate, and porous three-dimensional printed Ti cages), plating , and uncovertebrectomy (a technique of uncinate process resection) . The emergence of novel biologic therapies, including the use of mesenchymal stem cells and growth factors such as bone morphogenetic protein , has shown promise in promoting tissue regeneration and delaying degenerative progression, with some studies demonstrating significant improvements in patient-reported outcomes. However, the safety and long-term effectiveness of these techniques and biologic interventions continue to be subjects of ongoing investigation.

Study rationale and goals The field of surgical treatments for cervical degeneration is constantly evolving owing to advances in surgical techniques, biologic therapies, new emerging devices, and new diagnostic and evaluation tools, all with a keen focus on improving patient outcomes and minimizing complications. This dynamic field continues to drive advancements that hold the potential to enhance the quality of life for individuals affected by spinal degeneration. In view of this, under the AO CSH framework, the Cervical Mainstream study is dedicated to this field. AO CSH is a platform hosted by the AO Foundation for running clinical studies investigating similar diseases and/or patient groups in an efficient and effective manner.

Via the Cervical Mainstream, a large prospective multicenter patient cohort of cervical degenerative diseases who undergo anterior and/or posterior cervical fusion will be assembled. Key patient and treatment characteristics will be collected in a standardized manner. This patient cohort serves as a base for hypothesis generation, allowing the nesting of additional prospective or retrospective study(ies) within the running mainstream patient cohort and utilize its preexisting infrastructure, such as patient pool and data management resources.

Objectives Primary objective The primary objective is to form a large prospective multicenter patient cohort with standardized data collection of key patient and treatment characteristics that will drive hypothesis generation in patients with cervical degenerative diseases.

The mainstream study in AO Clinical Study Hub The current study also serves as the mainstream study of the AO CSH Cervical Mainstream. AO CSH is a platform hosted by the AO Foundation for running clinical studies investigating similar diseases and/or patient groups, eg, cervical degenerative diseases, in an efficient and effective manner. With the current study serves as the mainstream study, additional prospective or retrospective study(ies) can be nested to the AO CSH Cervical Mainstream. The process of "nesting" may involve identifying knowledge gap and generating hypothesis to be tested, which can be based on the exploratory analyses of the mainstream study data and identifying subgroups of patients within the mainstream study to form a study cohort for a hypothesis-testing study. An analogue to the CSH framework is the nested case-control study, a variation of a case-control study in which case and controls are drawn from a fully enumerated cohort [33]. Within the AO CSH framework, a prospective or retrospective study can be nested during the course of the mainstream study and utilizes its preexisting infrastructure, such as patient pool and data management resources. For example, the nested study can directly use the data fields already implemented in the mainstream study, provided that the same patient will be enrolled and consented to the mainstream study and the nested study(ies). Additional data fields that are needed for a nested study but not yet implemented in the mainstream study can always be developed for the specific nested study. The design and approach of AO CSH allows flexibility of adding different new prospective study(ies) over time while reducing the effort of recreating the same data fields and collecting the same data repeatedly.

In the AO CSH framework, this mainstream study may also drive further hypotheses and inform designs of future prospective studies to answer different research questions in specific subgroups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Undergoing primary surgical treatment for cervical degenerative disease
* Ability to provide informed consent according to the IRB/EC defined and approved procedures

Exclusion Criteria:

* Age under 18 years
* Patients with spinal infection
* Patients with spinal tumor
* Patients with acute spinal injuries/trauma within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cervical degenerative diseases undergoing primary anterior and/or posterior cervical fusion will be prospectively enrolled from participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2035-07-31 (Estimated)

PRIMARY OUTCOMES:
Form a large patient cohort | Baseline
  The primary objective is to form a large prospective multicenter patient cohort with standardized data collection of key patient and treatment characteristics that will drive hypothesis generation in patients with cervical degenerative diseases.